CLINICAL TRIAL: NCT03081026
Title: Transphyseal Vs. Physeal Sparing ACL Reconstruction in Skeletally Immature Patients: Risk of Subsequent Lower Extremity Growth Deformity
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Pro00063612
Record Dates: First submitted 2017-03-08; First posted 2017-03-15 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: ACL Reconstruction
Keywords: surgery; ages 6-16
MeSH Terms: interventions — Physical Examination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Ages less than 12: Those having ACL Reconstruction surgery during the desired dates at age 12 or less.
  Interventions: Diagnostic Test: Bilateral hip to ankle x-ray, exam and strength testing.
- Ages 12-13: Those having ACL Reconstruction surgery during the desired dates at ages 12 and 13.
  Interventions: Diagnostic Test: Bilateral hip to ankle x-ray, exam and strength testing.
- Ages 14 - 16: Those having ACL Reconstruction surgery during the desired dates at ages 14 - 16.
  Interventions: Diagnostic Test: Bilateral hip to ankle x-ray, exam and strength testing.

INTERVENTIONS:
Diagnostic Test: Bilateral hip to ankle x-ray, exam and strength testing. — Only an X-Ray is performed and reviewed to identify any growth disturbances.

SUMMARY:
To assess the risk of lower extremity angular growth deformity following anterior cruciate ligament (ACL) reconstructions in young patients who are not yet skeletally mature. The study will compare two surgical techniques (physeal sparing vs transphyseal).

DETAILED DESCRIPTION:
Background & Significance: In the adult population, the vast majority of ACL reconstructions are performed by drilling femoral and tibial bone tunnels. Because these patients have achieved physeal closure by the time of surgery, there is no risk of angular growth deformity when creating tibial and femoral tunnels. However, in the pediatric patient with open tibial and femoral physes, there is concern that drilling across the physes using standard tunnels may cause physeal injury with resultant angular deformity. Other surgical techniques have been described that allow the graft to be placed without drilling tunnels across the tibial and femoral physes but there is debate regarding whether or not these "physeal sparing" techniques are as effective as the transphyseal tunnel positions. Drilling the tunnels in the epiphysis to avoid the physis is a common "physeal sparing" technique. It is debated whether this technique could also cause growth disturbances. Given the increasing number of pediatric ACL injuries and that 95% of patients age 12 or less have open physes and that 94% of patients age 14 or greater have closed physes, this topic is of significant interest. Similar studies have been conducted but most have been either small and underpowered or have included older adolescent patients. At Duke Sports Sciences Institute, we have a sizable population of patients age 16 or less who have undergone ACL reconstruction with both transphyseal and all epiphyseal techniques. This provides a unique opportunity to analyze and compare these two groups with respect to clinical outcome and the incidence of growth disturbance or angular deformity

Design & Procedures: The investigator will conduct a review of medical records of seven providers at a single site institution to determine the subject population. Specifically, the investigator will look for patients who had an ACL reconstruction between the ages of 6-16 after January 1, 2005. The investigator will confirm in the medical record and in pre-operative radiographs that the growth plates were open at the time of surgery. Only subjects with open physeal will be enrolled in the study and they will be placed in 3 cohorts: Ages less than 12, 12-13, and 14 - 16. Subjects will be contacted by phone by a member of the team and asked to return to Duke Sports Sciences Institute to participate in the study. Upon arrival to clinic, subjects will be consented for the study and undergo a full physical exam - specifically targeting the gait and range of motion, as well as the Lachman, Anterior Drawer and Pivot Shift maneuvers to assess stability and functionality of the graft. In addition, they will complete a questionnaire designed to elicit patient satisfaction and level of activity/sports participation after the initial recovery period. Bilateral hip to ankle radiographs will be taken of each subject. These radiographs will be analyzed to assess for any angular deformity between the surgical and non-surgical leg. In addition, baseline knee x-rays will be reviewed for determination of skeletal maturity at time of injury/surgery. Data will be organized according to patients who underwent transphyseal reconstruction and patients who underwent physeal sparing reconstruction and separated into the corresponding age group. Comparisons will be made between the two surgical techniques based on the following criteria:

* Patient satisfaction and return to function
* Graft stability
* Angular deformity
* Skeletal maturity at the time of surgery

Study Interventions: Subjects will undergo physical examination (gait, inspections, range of motion and instability testing) and completion of an outcome tool survey (IKDC score/PediIKDC, VAS, Marx, and ACL-RSIsurvey). Subjects will undergo bilateral hip to ankle radiographic imaging to assess for growth deformity. Subjects will also be asked to give their permission to review their medical record and imaging pertinent to the knees and knee surgery.

Data Analysis & Statistical Considerations: Patient's data will be collected in a database program, indexed initially by medical record number. After case collection, case numbers will be applied and medical record numbers stripped from the data. The code linking medical record number to case number will be kept in a locked file with access limited to primary investigator.

Contingency analysis using the Fisher exact test will be used to compare the distribution of normal/nearly normal exam findings between the three cohorts

Descriptive statistics (mean, standard deviation and range) will be reported for each of these scores

Scores will be compared between the three cohorts using ANOVA with post-hoc analysis using Tukey's correction for multiple comparisons

Privacy, Data Storage & Confidentiality: The primary investigator will collect data in a computerized database using a commercially available database program. During collection, data will be indexed by the patient's medical record number. After data collection, a case number will be assigned to the data and the medical record number (the only identifying data collected) will be stripped from the database. The code linking medical record number to case number will be kept in a locked file with access limited to primary investigator. When the study is complete the code linking medical record numbers to case numbers will be destroyed. During data collection and review, protected health information will be available only to the primary investigator and will not be reused or disclosed to any other person or entity, except as required by law, for authorized oversight of the research study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be identified by reviewing medical records that include a procedure code for ACL reconstruction in patients between the ages of 6-16 at the time of surgery. Patients meeting the inclusion criteria will be contacted by phone and invited to participate in the study. A key personnel member who is part of the principal investigator's research staff will make phone contact with the patient. The study will be explained and any questions that the subject may have will be answered at that time. If the subject agrees to participate in the study, he/she will make an appointment at that time to come in to be consented and participate in the study and for imaging and testing at Duke Sports Sciences Institute.

Exclusion Criteria:

* Pregnant Females

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Single site patients of five orthopaedic sports medicine attendings who had an ACL reconstruction between the ages of 6-16 with open physes in the time interval from January 1, 2005-December 31, 2016.
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2020-03-06 (Actual); Study Completion 2020-03-06 (Actual)

PRIMARY OUTCOMES:
Limb length discrepancy | Clinic visit, approximately 1 hour
  Bilateral hip to ankle radiographs measurements.
Limb Angular alignment | Clinic visit, approximately 1 hour
  Bilateral hip to ankle radiographs measurements

SECONDARY OUTCOMES:
Range of motion measurements | Clinic visit, approximately 1 hour
  Each patient will be examined and measures of knee range of motion with a goniometer, Lachman and pivot shift will be performed. The Lachman and pivot shift will be dichotomized into two groups: normal/nearly normal and abnormal/severely abnormal.

OTHER OUTCOMES:
Patient Reported Outcomes surveys | Clinic visit, approximately 1 hour
  Pedi IKDC and level of activity/sports participation (UCLA Activity Score) after the initial recovery period.

CONTACTS AND LOCATIONS:
Overall Officials: Dean C Taylor, MD, Principal Investigator — Duke Sports Medicine
Locations (1):
- Duke Sports Science Institute, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
De-identified data will be sent to SmithNephew